CLINICAL TRIAL: NCT06850675
Title: Clinical Performance Comparison of the I-gel and Laryngeal Mask Airway-Supreme in Geriatric Patients: A Prospective Study
Brief Title: Comparison of Clinical Performance of Supraglottic Airway Devices
Acronym: SGADs
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nursen Karaca, Principal investigator, Ege University
Other Study IDs: 19-4.1T/40
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Supraglottic Airway Devices; Geriatric Patient
Keywords: supraglottic airway device; I-gel; LMA-Supreme; geriatric patients; clinical performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group ı-gel: The patients participating in the study were randomly assigned to two groups
  Interventions: Other: Clinical performance
- group lma-s: The patients participating in the study were randomly assigned to two groups
  Interventions: Other: Clinical performance

INTERVENTIONS:
Other: Clinical performance — Supraglottic airway devices were evaluated for ease of insertion, time of insertion, success rate at first attempt, number of attempts, ease of gastric tube insertion, oropharyngeal leak pressure, and intraoperative and postoperative complications

SUMMARY:
Abstract

Aim: To compare the clinical performance and pharyngolaryngeal complications of two second-generation, supraglottic airway devices (SGAD), the I-gel and Laryngeal Mask Airway-Supreme (LMA-Supreme), in geriatric patients undergoing elective surgery under general anesthesia.

Materials and Methods: After hospital ethics committee approval (19-4.1T/40- 17.04.2019) and written informed consent, patients aged 65 years and older, with an American Society of Anesthesiologists score of I-III, and who were scheduled for elective urological surgery under general anesthesia, were included prospectively. The patients were randomly divided into two equal sized groups, I-gel and LMA-supreme. The two groups were evaluated and compared for ease of supraglottic airway device insertion, time of insertion, success rate at first insertion, number of attempts, ease of gastric tube insertion, oropharyngeal leak pressure, and intraoperative and postoperative complications.

DETAILED DESCRIPTION:
After receiving approval from the Institutional Review Board (19-4.1T/40; 17.04.2019), patients aged 65 and older, who all had an American Society of Anesthesiologists (ASA) score of I-III, and who were scheduled for elective urological surgery under general anesthesia were prospectively recruited. Informed consent was obtained, either from the patients themselves or from a legal representative. Patients were excluded from the study if they were scheduled for emergency surgery, had unstable vital signs, a history of or suspicion of a difficult airway, preoperative sore throat, or a high risk of aspiration. The latter included individuals with a body mass index greater than 35 kg/m², gastroesophageal reflux, hiatal hernia, diabetic gastroparesis, or a history of medications affecting gastrointestinal motility. In addition, patients with a high risk of respiratory complications, such as those with asthma, chronic obstructive pulmonary disease, or recent pneumonia, abnormalities of the oral cavity or pharynx, cervical spine issues, communication difficulties, or those scheduled for surgeries lasting more than 90 minutes were also excluded.

The study took place from April 2019 to April 2020. The study included patients who were randomly assigned to two equally sized groups: the Laryngeal Mask Airway-Supreme (LMA-S) group and the I-gel group. This random assignment was conducted using a computer-assisted randomization method (www.randomizer.org). The insertion of the supraglottic airway device was performed by the same anesthesiologist, who had experience with at least 200 insertions of each type of supraglottic airway device and a first-attempt failure rate of less than 5% in a general patient population. During the procedure, patients were placed in the supine position with a standard pillow supporting their heads. Each device was prepared according to the manufacturer's recommendations, with the posterior and lateral sides lubricated using a water-soluble gel. The size of each device was selected based on the patient's weight, following the manufacturer's guidelines.

Upon the patient's admission to the operating room, standard monitoring was performed, which included non-invasive blood pressure (NIBP), pulse oximetry (SpO2), and electrocardiography (ECG). Preoxygenation was conducted for a minimum of three minutes using 100% oxygen at a fresh gas flow rate of 8 L/min. Anesthesia was induced intravenously with 1 mg/kg of 2% lidocaine, 1-2 µg/kg of fentanyl, and 2-3 mg/kg of propofol. No neuromuscular blocking agents were administered. The patients were manually ventilated with 100% oxygen and 2% sevoflurane until an adequate depth of anesthesia was achieved. This was determined by adequate jaw relaxation observed during the jaw thrust maneuver and the disappearance of the eyelash reflex. Once these criteria were met, the selected supraglottic airway device was inserted.

During the insertion of the I-gel, it was held by the bite block and advanced while the patient was in the "sniffing" position. This involved extending the head at the atlanto-occipital joint and flexing the neck while pushing the jaw downward. The device was directed towards the palate through the mouth and moved backward and downward until resistance was encountered.

During the insertion of the LMA-Supreme, the cuff was fully deflated first. The distal tip was then positioned against the inside of the upper teeth or gums. Using a slight crosswise approach, the device was gently slid inward, following the tongue, and advanced until resistance was felt. Once it was properly positioned, the cuff of the LMA-Supreme was inflated to a pressure of 60 cm H2O (measured with a VBM pressure gauge from Germany) and monitored regularly to maintain a constant cuff pressure. Adequate ventilation was verified through bilateral chest expansion, auscultation of lung sounds, and monitoring end-tidal CO2 (ETCO2) waveforms. If adequate ventilation was not achieved, the "jaw thrust maneuver" was attempted, along with neck extension or flexion, and made gentle adjustments to the position of the SGAD to ensure proper placement. Following successful placement, the patients were placed on a volume-controlled mode of mechanical ventilation using a mixture of 50%/50% oxygen and air. The tidal volume was set at 5-6 mL/kg, with a respiratory rate of 10-12 breaths per minute and an ETCO2 level maintained between 35-40 mmHg. Anesthesia was sustained with 1.0-2.0% sevoflurane in an oxygen/air mixture, along with an infusion of remifentanil at a rate of 0.25-0.5 µg/kg/min.

Oropharyngeal leak pressure (OLP) was measured during the operation after the SGAD was properly positioned. Measurements were taken at 15-minute intervals throughout the procedure and at the end of the surgery, just before removing the SGAD. OLP was determined by observing the pressure at which air leaked from the mouth, utilizing a fixed fresh gas flow of 5 L/min. The expiratory (APL) valve was closed at 30 cmH2O to ensure that the peak airway pressure did not exceed 40 cmH2O. The assessment of OLP used a five-point scale: 1=excellent (no air leak at 30 cmH2O); 2=good (air leak at 18-20 cmH2O); 3=moderate (air leak at 10-16 cmH2O); 4=poor (air leak at ≤ 8 cmH2O); and 5=placement/ventilation failure [16].

The placement time for the SGADs is defined as the duration between the removal of the face mask and the observation of the first ETCO2 waveform. The ease of insertion was evaluated using a 3-point scale: 1=easy (the device was placed successfully on the first attempt without resistance and without the need for additional maneuvers); 2=difficult (the device was placed on the first attempt with slight resistance, requiring either upward or downward movement of the device or lifting of the chin); or 3=very difficult (placement was only achieved on the second attempt despite maneuvers). In addition, the number of attempts and the ease of gastric tube insertion were assessed also using a 3-point scale after lubricating the gastric tube and advancing it through the gastric channel following SGAD placement: 1=first attempt (successful insertion on the first try); 2=second attempt (successful insertion on the second try); or 3=failure (insertion was not successful). Other recorded parameters included LMA-Supreme cuff pressure, operation duration (in minutes), anesthesia duration (in minutes), and intraoperative complications. The complications noted included dental, lip, and tongue injuries, hiccups, respiratory issues, such as desaturation SpO2 ≤ 92%, sudden increase in peak airway pressure, and/or changes in capnogram waveform, regurgitation/aspiration, laryngospasm, and apnea.

At the end of the operation, patients were given 1 mg/kg of tramadol and 10 mg/kg of paracetamol for pain management. The supraglottic airway device was removed once the patient demonstrated adequate spontaneous respiration and the ability to respond to verbal commands. During this process, any adverse events, such as laryngospasm, coughing, desaturation, and injuries to the tongue, teeth, or lips, as well as blood contamination on the laryngeal mask, were recorded. Patients were assessed for throat pain, hoarseness, and dysphagia at the second and twelfth hours postoperatively, with the symptoms graded as either present or absent.

Placing a supraglottic airway in patients undergoing surgery is a routine aspect of our anesthesia practices. The airway devices used in this study were standard for our procedures, and there were no non-routine applications performed on the patients included in the study. We only observed and recorded data from the patients.

ELIGIBILITY:
Inclusion criteria

* ≥65 age patients
* American Society of Anesthesiologists (ASA) score of I-III
* elective urological surgery

Exclusion Criteria:

* emergency surgery,
* unstable vital signs
* history of or suspicion of a difficult airway
* preoperative sore throat, or a high risk of aspiration
* body mass index ≥ 35 kg/m²
* gastroesophageal reflux
* hiatal hernia
* diabetic gastroparesis or a history of medications affecting gastrointestinal motility
* patients with a high risk of respiratory complications, such as those with asthma, chronic obstructive pulmonary disease, or recent pneumonia
* abnormalities of the oral cavity or pharynx,
* cervical spine issues,
* communication difficulties
* scheduled for surgeries lasting ≥ 90 minutes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 and older, who all had an American Society of Anesthesiologists (ASA) score of I-III, and who were scheduled for elective urological surgery under general anesthesia were prospectively recruited.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
The ease of insertion of supraglottic airway devices | intraoperative period
  The ease of insertion was evaluated using a 3-point scale: 1=easy (the device was placed successfully on the first attempt without resistance and without the need for additional maneuvers); 2=difficult (the device was placed on the first attempt with slight resistance, requiring either upward or downward movement of the device or lifting of the chin); or 3=very difficult (placement was only achieved on the second attempt despite maneuvers).
The time of insertion of supraglottic airway devices | intraoperative period
  The placement time for the supraglottic airway devices is defined as the duration between the removal of the face mask and the observation of the first end tidal carbon dioxide waveform
The ease of gastric tube insertion of supraglottic airway devices | intraoperative period
  The number of attempts and the ease of gastric tube insertion were assessed also using a 3-point scale after lubricating the gastric tube and advancing it through the gastric channel following SGAD placement: 1=first attempt (successful insertion on the first try); 2=second attempt (successful insertion on the second try); or 3=failure (insertion was not successful
oropharyngeal leak pressure of supraglottic airway devices | intraoperative period
  Oropharyngeal leak pressure (OLP) was measured during the operation after the SGAD was properly positioned. Measurements were taken at 15-minute intervals throughout the procedure and at the end of the surgery, just before removing the SGAD. OLP was determined by observing the pressure at which air leaked from the mouth, utilizing a fixed fresh gas flow of 5 L/min. The expiratory (APL) valve was closed at 30 cmH2O to ensure that the peak airway pressure did not exceed 40 cmH2O. The assessment of OLP used a five-point scale: 1=excellent (no air leak at 30 cmH2O); 2=good (air leak at 18-20 cmH2O); 3=moderate (air leak at 10-16 cmH2O); 4=poor (air leak at ≤ 8 cmH2O); and 5=placement/ventilation failure

SECONDARY OUTCOMES:
postoperative pharyngolaryngeal complications | up to postoperative 12 hour
  Patients were assessed for throat pain at the second and twelfth hours postoperatively, with the symptoms graded as either present or absent
postoperative pharyngolaryngeal complications | up to postoperative 12 hour
  Patients were assessed for hoarseness at the second and twelfth hours postoperatively, with the symptoms graded as either present or absent
postoperative pharyngolaryngeal complications | up to postoperative 12 hour
  Patients were assessed for dysphagia at the second and twelfth hours postoperatively, with the symptoms graded as either present or absent

CONTACTS AND LOCATIONS:
Overall Officials: NURSEN KARACA, MEDİCAL DOCTOR, Principal Investigator — Ege University Medical Faculty, Department of Anesthesiology and Reanimation
Locations (1):
- Ege University Medical Faculty Department of Anesthesiology and Reanimation, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I have not made a decision on this yet

REFERENCES:
- [Result] Kim EM, Kim MS, Koo BN, Lee JR, Lee YS, Lee JH. Clinical efficacy of the classic laryngeal mask airway in elderly patients: a comparison with young adult patients. Korean J Anesthesiol. 2015 Dec;68(6):568-74. doi: 10.4097/kjae.2015.68.6.568. Epub 2015 Nov 25. PMID 26634080
- [Result] Chen X, Jiao J, Cong X, Liu L, Wu X. A comparison of the performance of the I-gel vs. the LMA-Sduring anesthesia: a meta-analysis of randomized controlled trials. PLoS One. 2013 Aug 12;8(8):e71910. doi: 10.1371/journal.pone.0071910. eCollection 2013. PMID 23951266